CLINICAL TRIAL: NCT04847466
Title: A Phase II Study of Immunotherapy Combination: Irradiated PD-L1 CAR-NK Cells Plus Pembrolizumab Plus N-803 for Subjects With Recurrent/Metastatic Gastric or Head and Neck Cancer
Brief Title: Immunotherapy Combination: Irradiated PD-L1 CAR-NK Cells Plus Pembrolizumab Plus N-803 for Subjects With Recurrent/Metastatic Gastric or Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000096; 000096-C
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12-12

CONDITIONS: Gastroesophageal Junction (GEJ) Cancers; Advanced HNSCC
Keywords: PD-L1 t-haNK cells; GEJ cancer; Advanced HNSCC; Cellular Therapy; Keytruda
MeSH Terms: conditions — Neoplasms | interventions — ALT-803; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1 (Experimental): 1-week lead in for PD-L1 CAR NK cell monotherapy followed by combination therapy of Pembrolizumab plus N-803
  Interventions: Drug: N-803; Drug: Pembrolizumab; Biological: PD-L1 t-haNK

INTERVENTIONS:
Drug: N-803 — N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every 4 weeks (1 week after starting treatment with the PDL-1 CAR-NK cells).
Drug: Pembrolizumab — Pembrolizumab 400 mg will be administered as a 30-minute IV infusion every 6 weeks. Pembrolizumab will be administered on the same day as the PD-L1 CAR-NK cells.
Biological: PD-L1 t-haNK — PD-L1 CAR NK cells (2x109) will be administered by IV infusion over approximately 30 minutes every week. After the week 6 treatment, these cells will be given every 2 weeks.

SUMMARY:
Background:

Immunotherapy is a powerful tool in the fight against cancer. It uses the body s own immune system to fight the cancer. Unfortunately, cancer cells can find ways to escape from destruction by the body s immune system, even when immunotherapy is used.

Natural killer (NK) cells are an important part of the body s immune system and can help fight cancer. In combination with immunotherapy, researchers are using engineered NK cells that recognize and kill cancer cells trying to escape destruction by the immune system.

Objective:

To test the effectiveness of irradiated PD-L1 CAR-NK cells, combined with pembrolizumab and N-803, in people with advanced forms of gastric or head and neck cancer.

Eligibility:

Adults ages 18 and older with advanced gastric or head and neck cancer who have already had standard cancer treatment.

Design:

Participants will be screened with a medical history and physical exam. Their symptoms and ability to do normal activities will be assessed. They will have blood and urine tests. They will have imaging scans of the chest, abdomen, and pelvis.

Participants will get PD-L1 CAR-NK cells by intravenous (IV) infusion. They will get the cells once a week for 6 weeks. Then they will get the cells once every 2 weeks. Before each infusion, an IV catheter will be placed in a large arm vein for infusion of these treatments.

Participants will get pembrolizumab by IV every 6 weeks. They will get N-803 under the skin every 4 weeks.

Participants will get the study drugs for up to 2 years. They will have study visits every 1-2 weeks during treatment. They will have a safety visit 28 days after treatment ends.

After treatment ends, participants will be contacted for follow-up every 2 months for a year. Then they will be contacted every 6 months. They will have tumor scans every 6-12 weeks until their cancer gets worse.

DETAILED DESCRIPTION:
Background:

* Natural killer (NK) cells are an important component of an anti-tumor immune response.
* PD-L1 CAR-NK (PD-L1 t-haNKs) is an off the shelf, irradiated human, allogeneic, NK cell line that is frozen, shipped, thawed and then infused.
* PD-L1 CAR-NK cells have been engineered to have 3 adaptive modifications:

  * Expression of a chimeric antigen receptor (CAR) targeting the tumor-associated antigen PD-L1
  * Expression of the high-affinity variant (158V) of the human Fc gamma receptor (Fc gamma RIIIa/CD16a)
  * An endoplasmic reticulum-retained version of the human interleukin-2 (ERIL-2) cytokine.
* To improve the safety profile, PD-L1 CAR-NK cells are irradiated, thus inhibiting proliferation while maintaining cytotoxicity.
* Irradiated PD-L1 CAR-NK cells are highly effective at lysing PD-L1 expressing tumor cells as well as PD-L1 null tumor cells (via expression of native NK cell receptors).
* Preliminary clinical data from 10 participants treated with PD-L1 CAR-NK cells (NCT04050709) suggest PD-L1 CAR-NK are well tolerated at a dose of 2x10^9 cells intravenous (IV) twice per week. An additional 8 participants have received irradiated PDL1 CAR-NK under single patient INDs. PD-L1 CAR-NK cell treatment combined with PD-1 blockade and cytokine therapy may synergistically activate the T-cell and NK cell arms of the immune system and enhance anti-tumor activity.
* The combination of N-803 + PD-1/PD-L1 interaction blockade has a manageable safety profile

Objectives:

* Determine the 6-month progression free survival with irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab in participants with gastric/GEJ cancer.
* Determine the clinical response rate (CR+PR) with irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab in participants with Head and neck squamous cell carcinoma.

Eligibility:

* Gastric/GEJ cancer Cohort

  * Participants must have metastatic or unresectable locally advanced Gastric/GEJ cancer.
  * Participants must have evaluable disease with or without measurable disease by RECISTv1.1.
  * Participants must have completed, had disease progression on, or been ineligible to receive first-line systemic chemotherapy for advanced/metastatic disease and anti-PD-1 therapy for advanced/metastatic disease.
  * Participants with HER2 positive disease must have received HER2-targeted systemic therapy.
* Head and neck squamous cell carcinoma Cohort

  * Participants must have metastatic or unresectable locally advanced HNSCC.
  * Participants must have measurable disease by RECISTv1.1. If the participant is one of the first six participants enrolled on study and is part of the safety-lead in, either measurable or evaluable (e.g., ascites, elevated tumor marker, or lesion visualized on imaging) disease will be permitted.
  * Participants must have received or been ineligible to receive first-line systemic chemotherapy and must have received systemic anti-PD-1 therapy (in the first-line or subsequent-line setting).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Age >= 18 years

Design:

* This is an open label, single center, phase II trial using a safety lead-in to assess the safety and tolerability of irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab in participants with head and neck squamous cell carcinoma and/or gastric/GEJ cancer.
* The phase II objectives of this study is to assess 6-month progression free survival (PFS) and clinical response rate (CR+PR) in participants with gastric/GEJ cancer and head and neck squamous cell carcinoma, respectively.
* Participants will enroll and receive 1 dose of PD-L1 CAR-NK cell monotherapy (week -1) for PK/PD studies before starting the combined treatment of Pembrolizumab and N-803 one week later (week 0). PD-L1 CAR-NK cells (2x10^9) will be given intravenously every week until week 6 and then every two weeks from 6 week onward.
* The accrual is 50 evaluable participants. To allow for a small number of inevaluable participants, the accrual ceiling will be set at 55 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Gastric/GEJ cancer Cohort:

  * Participants must have metastatic or unresectable locally advanced Gastric/GEJ cancer that has been histologically confirmed.
  * Participants must have radiologically evaluable disease, with or without measurable lesions by RECISTv1.1. Evaluable but non-measurable disease include small lesions (longest diameter <10mm or pathological lymph nodes with >=10 to <15mm short axis), ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.
  * Participants must have received or been ineligible to receive first line systemic chemotherapy for Gastric/GEJ cancer. Participants with HER2 positive disease must have received HER2-targeted therapy.
* Head and neck squamous cell carcinoma Cohort

  * Participants must have metastatic or unresectable locally advanced HNSCC that has been histologically confirmed.
  * Participants must have measurable disease by RECISTv1.1. If the participant is one of the first six participants enrolled on study and is part of the safety-lead in, either measurable or evaluable (e.g. ascites, elevated tumor marker, or lesion visualized on imaging) disease will be permitted.
  * Participants must have received or been ineligible to receive first-line systemic chemotherapy and must have received systemic anti-PD-1 therapy (in the first-line or subsequent-line setting).
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of this investigation combination therapy in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status <2 (Karnofsky >60%)
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL
  * platelets >=100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal
  * creatinine Creatinine within 1.5X upper limit of normal institutional limits
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first 7 weeks of therapy.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants on therapeutic anticoagulation with warfarin must have an international normalized ratio (INR) that is within target range for their condition at the time of enrollment.
* The effects of PD-L1 t-haNKs with N-803 and pembrolizumab on the developing human fetus are unknown. For this reason and because these investigational agents teratogenicity is unknown, individuals of child-bearing potential and individuals who can father a child must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation and for at least 4 months after last dose of study drug pembrolizumab.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents or concurrent anticancer treatment. Palliative radiotherapy is allowed.
* Participants with concurrent use of systemic steroids (within 10 days of enrollment), except for physiologic doses of systemic steroid replacement or local (topical, nasal, intraarticular or inhaled) steroid use.
* Participants with active systemic autoimmune disease (e.g., lupus erythematosus, rheumatoid arthritis, Addison s disease, autoimmune disease associated with lymphoma, inflammatory bowel disease). Participants with autoimmune endocrine disorders controlled with medical management (e.g. thyroid disorders, type 1 diabetes, or adrenal insufficiency) will not be excluded
* Participants with a history of grade 3 or higher immune-related adverse events attributed to pembrolizumab or other anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy. This exclusion does not apply to participants with permanent endocrine insufficiencies (e.g. adrenal insufficiency or hypothyroidism) under satisfactory medical management. Additionally, participants with grade 2 adverse events attributed to these classes of agents will be excluded with the exception of rash, transient hyperthyroidism, transient liver enzyme abnormalities or other transient events that resolved without steroids or immunomodulatory agents.
* HIV or HBV infection due to unknown effect of PD-L1 targeting via a CAR or N-803 in these chronic viral infections.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled serious cardiac arrhythmia, clinically significant coagulopathy or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant individuals are excluded from this study because PD-L1 targeting via a CAR has unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PD-L1 targeting via a CAR and N-803, nursing should be discontinued if the mother is treated on this study for the duration of study participation and for at least 4 months after last dose of any study drug.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the clinical response rate (CR+PR) with irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab in patients with head and neck squamous cell carcinoma and gastric/GEJ cancer. | every 6 weeks
  Clinical response rate (CR+PR)

SECONDARY OUTCOMES:
To assess the progression free survival (PFS) in patients with HNSCC and/or gastric/GEJ cancer treated with irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab | Until progression or death
  The proportion of patients that have progressive disease after 18 months
To assess the safety and tolerability of irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab in patients with head and neck squamous cell carcinoma and/or gastric/GEJ cancer | 28 days after treatment (Study Calendar-Last AE evaluation)
  List of adverse event frequency
To assess duration of response in patients with HNSCC and/or gastric/GEJ cancer treated with irradiated PD-L1 CAR-NK cells in combination with N-803 plus pembrolizumab | Until progression or death
  The time when the proportion of patient's tumors shrunk after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000096-C.html